CLINICAL TRIAL: NCT00012766
Title: Effectiveness of Team Treatment of Depression in Primary Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 95-097
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-12

CONDITIONS: Depression; Primary Health Care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Integrated team care

INTERVENTIONS:
Behavioral: Integrated team care

SUMMARY:
Most depression treatment takes place in primary care, where the condition continues to be under-detected and under-treated. A collaborative care model derived from chronic illness management theory has been successful in improving care in other managed care settings.

DETAILED DESCRIPTION:
Background:

Most depression treatment takes place in primary care, where the condition continues to be under-detected and under-treated. A collaborative care model derived from chronic illness management theory has been successful in improving care in other managed care settings.

Objectives:

This effectiveness study adapted collaborative care to the VA primary care setting ("collaborative care") and compared it with consult-liaison care ("CL care").

Methods:

Patients within a VA primary care clinic were randomly assigned by firm to the two interventions.

In collaborative care, existing staff resources were reorganized to form a multidisciplinary mental health specialist team. The team developed a treatment plan based on an initial assessment and suggested the plan to the primary care provider. Primary care providers' treatment efforts were then supported by brief Social Work telephone calls designed to support adherence and monitor symptomatology. Treatment results were systematically reviewed and suggestions for treatment modification were fed back to the primary providers. In CL care, the primary care providers were informed of the diagnosis and study clinicians facilitated referrals to Psychiatry residents in-clinic as requested. Mailed and in-clinic surveys and provider referral were used to recruit 168 collaborative care and 186 CL care patients who met criteria for major depression and/or dysthymia based on structured interview. Patients were excluded only if they required immediate inpatient care, had a pending mental health specialty clinic appointment, or had primary alcohol abuse. Outcome data on the SCL-20 depression symptomatology measure, Veterans SF-36, and Sheehan Disability Scale were collected at baseline, 3 and 9 months. VA utilization and costs of care were analyzed.

Status:

Complete. Final Report submitted June 30, 2001.

ELIGIBILITY:
Inclusion Criteria:

Several screening methods including mailed and in-clinic surveys and provider referral were used to recruit 168 team and 188 CL study patients who met criteria for major depression and/or dysthymia based on structured interview. Patients were excluded only if they required immediate inpatient care, had a pending mental health specialty clinic appointment, had primary alcohol abuse, or were too impaired to participate in the screening interview. Outcome data on the SCL-20 depression symptomatology measure, SF-36V, and Sheehan functional impairment measure were collected at baseline, 3 and 9 months.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan C. Hedrick, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Edmund F. Chaney, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

REFERENCES:
- [Result] Hedrick SC, Chaney EF, Felker B, Liu CF, Hasenberg N, Heagerty P, Buchanan J, Bagala R, Greenberg D, Paden G, Fihn SD, Katon W. Effectiveness of collaborative care depression treatment in Veterans' Affairs primary care. J Gen Intern Med. 2003 Jan;18(1):9-16. doi: 10.1046/j.1525-1497.2003.11109.x. PMID 12534758
- [Result] Liu CF, Hedrick SC, Chaney EF, Heagerty P, Felker B, Hasenberg N, Fihn S, Katon W. Cost-effectiveness of collaborative care for depression in a primary care veteran population. Psychiatr Serv. 2003 May;54(5):698-704. doi: 10.1176/appi.ps.54.5.698. PMID 12719501
- [Result] Fischer EP, Marder SR, Smith GR, Owen RR, Rubenstein L, Hedrick SC, Curran GM. Quality Enhancement Research Initiative in Mental Health. Med Care. 2000 Jun;38(6 Suppl 1):I70-81. doi: 10.1097/00005650-200006001-00008. PMID 10843272
- [Result] Felker BL, Hedrick SC, Chaney EF, Liu CF, Heagerty P, Caples H, Lin P, Katon W. Identifying Depressed Patients With a High Risk of Comorbid Anxiety in Primary Care. Prim Care Companion J Clin Psychiatry. 2003 Jun;5(3):104-110. doi: 10.4088/pcc.v05n0301. PMID 15154020
- [Result] Lin P, Campbell DG, Chaney EF, Liu CF, Heagerty P, Felker BL, Hedrick SC. The influence of patient preference on depression treatment in primary care. Ann Behav Med. 2005 Oct;30(2):164-73. doi: 10.1207/s15324796abm3002_9. PMID 16173913
- [Result] Kanter JW, Epler AJ, Chaney EF, Liu CF, Heagerty P, Lin P, Felker B, Hedrick SC. Comparison of 3 Depression Screening Methods and Provider Referral in a Veterans Affairs Primary Care Clinic. Prim Care Companion J Clin Psychiatry. 2003 Dec;5(6):245-250. doi: 10.4088/pcc.v05n0601. PMID 15213794